CLINICAL TRIAL: NCT04794530
Title: COCOA Flavanols to Improve Walking Performance in PAD: the COCOA-PAD II Trial
Brief Title: The COCOA-PAD II Trial
Acronym: COCOA-PAD II
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Minnesota (Other); University of Chicago (Other)
Responsible Party: Principal Investigator, Mary McDermott, Jeremiah Stamler Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00213897; R01AG068458-01A1 (NIH)
Record Dates: First submitted 2021-03-07; First posted 2021-03-12 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Peripheral Artery Disease
Keywords: cocoa flavanols
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- cocoa flavanols (Active Comparator)
  Interventions: Drug: cocoa flavanols
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: cocoa flavanols — The cocoa flavanols intervention is manufactured by Mars Inc. Participants randomized to cocoa flavanols will take two capsules daily of cocoa flavanols. The two capsules of cocoa flavanols will contain approximately 500 mg of cocoa flavanols and appoximately 80 mg of (-)-epicatechin.
  Arms: cocoa flavanols
Drug: placebo — The placebo intervention will be manufactured by Mars Inc. and will appear identical to the cocoa flavanols intervention. Participants will take two capsules daily of placebo. The placebo will be a cellulose based capsule and will not contain cocoa flavanols or (-)-epicatechin.
  Arms: placebo

SUMMARY:
Among people with peripheral artery disease (PAD) age 55 and older, the investigators will test the hypothesis that PAD participants randomized to cocoa flavanols will have greater improvement or less decline in six-minute walk distance at six-month follow-up, compared to those randomized to placebo. The study will randomize 190 participants with PAD age 55 and older to one of two groups for six months: cocoa flavanols vs placebo. Our primary outcome is change in six-minute walk distance at six-month follow-up. Secondary outcomes are Actigraph-measured physical activity, brachial artery flow-mediated dilation (FMD), gastrocnemius muscle biopsy measures of endothelial nitric oxide synthase (eNOS) and phosphorylated eNOS, gastrocnemius muscle perfusion (measured by magnetic resonance imaging (MRI)) and gastrocnemius muscle characteristics (measured by muscle biopsy).

To achieve the specific aims, the study will randomize 190 participants age 55 and older with PAD to one of two groups: cocoa flavanols vs placebo. Participants will be followed for six months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55 and older
2. Presence of peripheral artery disease (PAD). PAD will be defined as either:

   1. An ABI <= 0.90 at baseline.
   2. Vascular lab evidence of PAD (such as a toe brachial pressure < 0.70 or an ankle brachial index less than or equal to 0.90), or angiographic evidence of PAD defined as at least 70% stenosis of an artery supplying the lower extremities.
   3. An ABI of >0.90 and <=1.00 who experience a a 20% or greater drop in ABI in either leg after the heel-rise test will also be included.

Exclusion Criteria:

1. Above- or below-knee amputation
2. Critical limb ischemia
3. Wheelchair confinement or requiring a walker to ambulate
4. Walking is limited by a symptom other than PAD
5. Current foot ulcer on bottom of foot
6. Failure to successfully complete the one-week study run-in
7. Planned major surgery, coronary or leg revascularization during the next eight months
8. Major surgery, coronary or leg revascularization or major cardiovascular event in the previous three months
9. Major medical illness including lung disease requiring oxygen, Parkinson's disease, a life-threatening illness with life expectancy less than eight months, or cancer requiring treatment in the previous two years. [NOTE: potential participants may still qualify if they have had treatment for an early stage cancer in the past two years and the prognosis is excellent. Participants who require oxygen only at night may still qualify.]
10. Mini-Mental Status Examination (MMSE) score < 23
11. Allergy to the study intervention
12. Potential participants who have taken cocoa supplements in previous three months, are unwilling to avoid taking cocoa flavanol supplements, or are consuming dark chocolate regularly (i.e. approximately 1.5 ounces of dark chocolate more than three times per week, or more than 4.5 ounces per week).
13. Non-English speaking
14. Participation in or completion of a clinical trial in the previous three months. [NOTE: after completing a stem cell or gene therapy intervention, participants will become eligible after the final study follow-up visit of the stem cell or gene therapy study so long as at least six months have passed since the final intervention administration. After completing a supplement or drug therapy (other than stem cell or gene therapy), participants will be eligible after the final study follow-up visit as long as at least three months have passed since the final intervention of the trial.]
15. Visual impairment that limits walking ability
16. Six-minute walk distance of <500 feet or >1600 feet.
17. Participation in a supervised treadmill exercise program in previous three months
18. Unable to tolerate caffeine
19. In addition to the above criteria, investigator discretion will be used to determine if the trial is unsafe or not a good fit for the potential participant

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2021-11-19 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Six-month change in six-minute walk distance | Baseline to six-month follow-up
  Change in six-minute walk distance at six-month follow-up will be compared between those randomized to cocoa flavanols vs. those randomized to placebo.

SECONDARY OUTCOMES:
Six-month change in gastrocnemius muscle perfusion (measured by magnetic resonance imaging (MRI)) | Baseline to six-month follow-up
  Change in gastrocnemius muscle perfusion (measured by MRI) at six-month follow-up will be compared between those randomized to cocoa flavanols vs. those randomized to placebo.
Six-month change in brachial artery flow-mediated dilation (FMD) | Baseline to six-month follow-up
  Change in brachial artery flow-mediated dilation (FMD) at six-month follow-up will be compared between those randomized to cocoa flavanols vs. those randomized to placebo.
Six-month change in Actigraph-measured physical activity | Baseline to six-month follow-up
  Change in Actigraph-measured physical activity at six-month follow-up will be compared between those randomized to cocoa flavanols vs. those randomized to placebo.
Six-month change in calf muscle endothelial nitric oxide synthase (eNOS) and phosphorylated eNOS | Baseline to six-month follow-up
  Change in calf muscle biopsy measures of eNOS and phosphorylated eNOS at six-month follow-up will be compared between those randomized to cocoa flavanols vs. those randomized to placebo.
Six-month change in calf muscle characteristics (measured by calf muscle biopsy) | Baseline to six-month follow-up
  Change in calf muscle characteristics (measured by calf muscle biopsy) at six-month follow-up will be compared between those randomized to cocoa flavanols vs. those randomized to placebo.
Six minute walk at two and four week follow-up after intervention completion. | Six-month follow-up to 2- and 4-weeks post follow-up
  The trial will determine whether cocoa flavanols, compared to placebo, have a persistent effect on improved six-minute walk distance at two weeks and four weeks after the study intervention is completed

OTHER OUTCOMES:
Six-month change in plasma abundance of cocoa flavanols | Baseline to six-month follow-up
  The trial will determine whether lower plasma abundance of cocoa flavanols at baseline and whether greater increases in plasma abundance of cocoa flavanols at 6-month follow-up are associated with greater improvement in six-minute walk distance at 6-month follow-up, compared to higher plasma abundance of cocoa flavanols at baseline and compared to smaller increases in plasma cocoa flavanols at 6-month follow-up, respectively
Association of calf perfusion with baseline gut microbial diversity with response to cocoa flavanols | Baseline to six-month follow-up
  The trial will determine whether baseline gut microbial diversity and composition are associated with the degree of response to cocoa flavanols, compared to placebo, measured by greater improvement calf perfusion at 6-month follow-up.
Association of six-minute walk distance with baseline gut microbial diversity with response to cocoa flavanols | Baseline to six-month follow-up
  The trial will determine whether baseline gut microbial diversity and composition are associated with the degree of response to cocoa flavanols, compared to placebo, measured by greater improvement in six-minute walk distance at 6-month follow-up.
Six-month change in gut microbial diversity | Baseline to six-month follow-up
  The trial will determine whether cocoa flavanols, compared to placebo, favorably alter gut microbial diversity at six-month follow-up.
Six-month change in gut microbial composition | Baseline to six-month follow-up
  The trial will determine whether cocoa flavanols, compared to placebo, favorably alter gut microbial composition at six-month follow-up.
Association of six-minute walk distance with six-month change in gut microbial composition | Baseline to six-month follow-up
  The trial will determine whether cocoa flavanol-induced changes in gut microbial composition, compared to placebo, between baseline and 6-month follow-up are associated with greater improvement in six-minute walk distance.
Association of calf perfusion with six-month change in gut microbial composition | Baseline to six-month follow-up
  The trial will determine whether cocoa flavanol-induced changes in gut microbial composition, compared to placebo, between baseline and 6-month follow-up are associated with greater improvement in calf perfusion.
Association of metabolomic profiles with improved six-minute walk distance. | Baseline to six-month follow-up
  The trial will perform microbe-associated metabolomic profiling in blood and stool at six-month follow-up to identify metabolomic profiles that are associated with improved six-minute walk distance at 6-month follow-up.
Association of metabolomic profiles with improved calf perfusion | Baseline to six-month follow-up
  The trial will perform microbe-associated metabolomic profiling in blood and stool at six-month follow-up to identify metabolomic profiles that are associated with improved calf perfusion at 6-month follow-up.
Association of metabolomic profiles with six-minute walk distance | Baseline to six-month follow-up
  The trial will perform microbe-associated metabolomic profiling in blood and stool at six-month follow-up to identify metabolomic profiles that are associated with improved six-minute walk distance at six-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Mary McDermott, MD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No